CLINICAL TRIAL: NCT06277726
Title: The Effect of Emotional Freedom Technique and Music Recital on Pain and Anxiety Experienced During Intrauterine Device Application
Brief Title: The Effect of Two Non-pharmacological Methods on Pain and Anxiety Experienced During Intrauterine Device Application.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ceylan Guzel Inal, Lecturer, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IU-SBE-CGI-01
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Intrauterine Devices
Keywords: intrauterine device; pain; anxiety; emotional freedom technique; music; nursing
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled study with pre-test post-test group
Who Masked: Participant, Investigator
Masking Description: In order to ensure randomization and prevent contamination between groups, data will be collected in a sequence such that emotional freedom technique is collected one week, music is collected one week, and control group data is collected one week. It will be decided by drawing lots which group's data will be collected first.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional freedom technique group (Experimental): Pre-test data will be collected after women are informed about the emotional freedom technique. After the pre-test data is collected, the emotional liberation technique will be applied to the women. After the emotional liberation technique session is completed, the intrauterine device (IUD) will be applied. Post-test data will be collected within 10 minutes after IUD application is completed.
  Interventions: Other: Emotional freedom technique group
- Music group (Experimental): Women in the music group will be informed about the procedure steps before intrauterine device (IUD) application and pre-test data will be collected. After the pre-test data is collected, the music list prepared by the women and researchers will be shown and the women will be asked to choose a piece. Women who do not want to listen to any music on this list will be allowed to listen to the music they prefer. The music concert will be performed with headphones, and women will be asked to listen to the music until the IUD application process is completed. Post-test data will be collected within 10 minutes after IUD application.
  Interventions: Other: Music group
- Control group (Other): No intervention will be applied to women in the control group.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Emotional freedom technique group — Emotional freedom technique will be applied to women in this group before intrauterine device application.
  Arms: Emotional freedom technique group
Other: Music group — Women in this group will wear headphones and listen to music throughout the intrauterine device application.
  Arms: Music group
Other: Control group — No intervention will be applied to women in the control group.
  Arms: Control group

SUMMARY:
The purpose of this study is to determine the effect of emotional freedom technique and music, which are effective in relieving pain and anxiety, on the pain and anxiety that occur during intrauterine device application.

DETAILED DESCRIPTION:
Intrauterine devices, which are considered one of the most effective contraceptive methods, can be effective up to 99% when used correctly. While 17% of women of reproductive age around the world use intrauterine devices, 13.7% of women in our country prefer intrauterine devices as a contraceptive method. Intrauterine devices have many benefits such as being easy to use, returning fertility when removed, being able to be used for a long time, and being low in cost. Intrauterine devices are recommended to women as the first choice by medical institutions due to their high effectiveness rates. However, anxiety and pain experienced during the intrauterine device placement procedure may prevent women from choosing intrauterine devices as a birth control method. Music and emotional liberation techniques can be used as alternative methods to relieve pain and anxiety. In this research, the effects of emotional freedom technique and music, which are effective on pain and anxiety, on pain and anxiety during intrauterine device application will be investigated. Additionally, it will be tested whether the emotional liberation technique and music are superior to each other in relieving the pain and anxiety that occur during intrauterine device application. Additionally, no research has been found in the literature examining the effects of emotional liberation technique and music recital on the pain and anxiety experienced during intrauterine device application. With this research, the gap in the field will be eliminated and new research and applications will be structured.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreeing to participate in the research
* Being between the ages of 18-49

Exclusion Criteria:

* Having a verbal communication problem
* Being medically diagnosed with a psychiatric disorder
* Presence of wounds, scars and infections in the areas touched in the emotional freedom technique
* Having a hearing problem
* Having had an intrauterine device (IUD) inserted before
* Being exposed to domestic violence
* Being diagnosed with any medical condition (hypertension, diabetes, etc.)
* Having used analgesics seven hours before the procedure
* Having a gynecological examination just before IUD application

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 168 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | It will be used for 10 months, which is the data collection period. It will be used before and ten minutes after intrauterine device application.
  A visual analog scale will be used to measure the pain caused by intrauterine device application. It is a two-ended scale that is used to measure the intensity of pain and is graded on a horizontal line, with one end starting from 0 and the other end ending at 10. The patient is asked to mark a point on this line that corresponds to the intensity of pain he feels. The numerical value marked by the patient indicates the severity of pain. A VAS value of 0 indicates no pain, 1-3 indicates mild pain, 4-6 indicates moderate pain, 7-9 indicates severe pain, and 10 indicates unbearable pain.
State Anxiety Inventory | It will be used for 10 months, which is the data collection period. It will be used before and ten minutes after intrauterine device application.
  State anxiety inventory; It is a scale consisting of 20 questions that include the options of (1) not at all, (2) a little, (3) quite a bit, (4) completely, depending on the severity of the emotions at that moment, so that the individual can describe how he feels at a certain moment. Accordingly, the total score obtained from the scale can vary between 20 and 80. A high score from the scale indicates a high level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ceylan GÜZEL İNAL, Lecturer, Principal Investigator — Şırnak Universty; Sermin TİMUR TAŞHAN, Prof. Dr., Study Director — İnönü Universty
Locations (1):
- Şırnak State Hospital, Şırnak, Turkey (Türkiye)